CLINICAL TRIAL: NCT05127031
Title: Validity and Reliability of VO2-max Measurements in Persons With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: RHP21
Record Dates: First submitted 2021-10-27; First posted 2021-11-19 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2021-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — A blood lactate test would be completed immediately after the VO2-max test.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Each participant would complete four test days and each test day is separated by 7-10 days. At each test day the participants would complete a graded maximal exercise test (VO2max-test), a chair rise (Linear encoder) as well as measuring of basic demographic outcomes (weight, fat%,blood pressure etc.). The first test day would further include a motor (MDS-UPDRS III) and cognitive examination (MoCA), a questionnaire about quality of life (PDQ-39) and one about depression (BDI-II). Furthermore, the first test day would include two test of walking performance (6 minutes walk test and Time Up and Go). Two of the test days would be completed while the participants are off their Parkinson disease medication for at least 12 hours, while the other two test days would be completed while on their Parkinson medication. The order of the tests would be randomized. It is hypothesized that the VO2max test would be reliable and valid when participants are on medication, while off-medication would affect the reliability and validity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 year
* Written informed consent
* Diagnosed with idiopathic Parkinson's disease
* Hoehn & Yahr ≤ 3
* Taking dopaminergic medication
* Able to complete a maximal aerobic test on a bicycle

Exclusion Criteria:

* Dementia
* Alcohol abuse
* Pacemaker
* Serious cardiovascular, respiratory, orthopedic or other comorbidities excluding maximal exercise participation.
* Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is selected from hospitals in Denmark, including Aarhus University Hospital, Lillebælt Hospital and Odense University Hospital. Moreover, the population is also selected from private neurological clinics in Esbjerg, Viborg, Aarhus and Skanderborg. In addition, the study population is recruited via the Danish Parkinson's disease association (including their Facebook website).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
VO2max (O2ml/min/kg) change | Up to 40 days
  The maximal oxygen consumption during and graded exercise test. Used to asses the day to day variation between two test.
VO2 plateau (Primary validity criterion) | Up to 40 days
  Looking at the difference between the actual measure of VO2 at the end of the VO2-max test and the predicted VO2 calculated using a linear regression.
Respiratory exchange ratio (RER) (secondary validity criterion) | Up to 40 days
  The ratio between VCO2 (L/min) and VO2 (L/min)
Blood lactate (secondary validity criterion) | Up to 40 days
  Blood lactate level taken from a fingertip one minute after the VO2max has ended.
Maximal heart rate (beats/min) (secondary validity criterion) | Up to 40 days
  We would detect the maximal heart rate at the end of the test
Rating perceived exertion (RPE) (secondary validity criterion) | Up to 40 days
  Using the Borg scala, we would determine the RPE at the end of the test.

SECONDARY OUTCOMES:
Chair rise - maximal power output (W) change | Up to 40 days
  The maximal power output measured during af chair rise (Linear Encoder). Using the change between two tests to evaluate the reliability
Parkinson's Disease Questionnaire (PDQ-39) | At the first test day
  A questionnaire to evaluate the quality of life with scores ranging from 0-100 (higher scores indicating worse quality of life)
Beck Depression Inventory-II (BDI-II) | At the first test day
  To evaluate depression. Scores ranges from 0-63 with higher scores indicating more severe depressive symptoms
Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating scale (MDS-UPDRS) III | At the first test day
  A motor examination done by an educated assessor. Scores ranges from 0-132 with higher scores indicating more severe motor disability.
6-minute walk test (6MWT) | At the first test day
  To measure the distance, the participant is able to walk over 6 minutes using a 30 meter track.
Timed up and go (TUG) | At the first test day
  Participants have to rise from a chair, walk three meters and go back and sit on the chair again as fast as possible, without running
The Montreal Cognitive Assessment (MoCA) | At the first test day
  Participants have to complete different task using the MoCA.
Weight (kg) | Four times (one at each visit) during af 40 days period
  We would collect information about weight using bioimpedance sensor (TANITA SC220).
Blood pressure (systolic/diastolic) (mmHg) | Four times (one at each visit) during af 40 days period
  Using a blood pressure monitor to ensure that participants do not have a blood pressure above 160/110 mmHg at test day.
Date of diagnosis (month and year) | At first visit only
  Collecting information from when participants were diagnosed with Parkinson disease to detect disease duration (years)
Medication | At first visit only
  We want to know what type of medication that they use to ensure that participants fulfill the inclusion criterion

CONTACTS AND LOCATIONS:
Locations (1):
- Sport Science, Department of Public Health, Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No